CLINICAL TRIAL: NCT06326918
Title: The Difference of Duodenal Microbiota Between Patients With Functional Dyspepsia and Control: a Pilot Study
Brief Title: Duodenal Microbiota in Functional Dyspepsia
Status: Recruiting | Type: Observational
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Associate Professor, King Chulalongkorn Memorial Hospital
Other Study IDs: RP026
Record Dates: First submitted 2024-03-18; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Functional Dyspepsia
Keywords: Duodenal microbiota; Gut microbiome; Functional dyspepsia; Next generation sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Duodenal mucosa by duodenal mucosal brushing and duodenal mucosal biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Functional dyspepsia: 1. Patients who are 18 years old or more and exhibit at least one of the following four symptoms for the last 3 months, with symptom onset occurring at least 6 months prior to diagnosis.
     1.1 Postprandial distress syndrome (symptoms occurring at least 3 days per week), including:
     * Postprandial fullness and/or
     * Early satiation
     1.2 Epigastric pain syndrome (symptoms occurring at least 1 day per week), including:
     * Epigastric pain and/or
     * Epigastric burning
  2. Participants undergo esophago-gastro duodenoscopy (EGD) to confirm the absence of any structural abnormalities.
  Interventions: Diagnostic Test: Duodenal mucosal brushing; Diagnostic Test: Duodenal mucosal biopsy
- Control: * Patients with no or minimal upper GI symptoms (not match the criteria of FD) and current EGD appear normal or insignificant gastritis
  * Age- and sex-matched to the functional dyspepsia (FD) patient group.
  Interventions: Diagnostic Test: Duodenal mucosal brushing; Diagnostic Test: Duodenal mucosal biopsy

INTERVENTIONS:
Diagnostic Test: Duodenal mucosal brushing — Duodenal mucosal brushing will be performed at duodenal bulb.
Diagnostic Test: Duodenal mucosal biopsy — Duodenal mucosal biopsy will be performed at duodenal bulb.

SUMMARY:
The goal of this observational study is to assess the type of duodenal microbiota and duodenal microbiome in in FD patients compared to control group. The main questions it aims to answer are:

* What are the differences in the type of duodenal microbiota and is there a difference in duodenal microbiome diversity between patients diagnosed with functional dyspepsia (FD) and the control group?
* Are there any significant variations in the composition and diversity of gut microbiota between patients with FD and the control group, considering the method of sample collection (duodenal brushing vs. duodenal biopsy)?

DETAILED DESCRIPTION:
Dyspepsia, a common GI disorder, affects a significant portion of the global population, with a prevalence as high as 66% in Thailand. Functional dyspepsia (FD) is characterized by no detectable structural abnormalities during endoscopic examinations and significantly impacts health-related quality of life. Dysregulation of the gut-brain axis is hypothesized to contribute to motility disorders, visceral hypersensitivity, and mucosal/immune function changes in FD.

Recent studies have characterized the microbiota of the duodenal mucosal-associated microbiome (MAM) in patients with functional dyspepsia (FD). However, duodenal microbiota in FD patients compared to healthy control remains unclear with conflicting results. The number of studies evaluating this is limited, and a well-designed study comparing the duodenal microbiota of patients with functional dyspepsia to control group will advance our understanding of the potential role of the microbiome in FD. Therefore, the aim of this study is to compare the duodenal microbiota of patients with FD and those without upper GI symptoms.

This study is pilot phase, cross-sectional and case-control study that aims to evaluate microbiota profile in patients with functional dyspepsia, compared to those without functional dyspepsia by using mucosal brush sampling and mucosal biopsy sampling.

Study protocol include Age, gender, BMI, smoking history, history of PPI use within 2 weeks, history of antibiotic use within 4 weeks, history of probiotic use within 4 weeks will be recorded in case record form.

After consent, standard EGD will be performed. The duodenal mucosa using mucosal brushing with sterile sheathed brush, duodenal mucosal biopsy by standard forceps biopsy will be done respectively. ㆍ The duodenal mucosal specimen will be keep in sterile tube and immediate keep in freezing at -80C (allow room temperature <2 hr) for 16sRNA sequencing analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Functional dyspepsia group 1.1 Patients who are 18 years old or more and exhibit at least one of the following four symptoms for the last 3 months, with symptom onset occurring at least 6 months prior to diagnosis.

   1.1.1 Postprandial distress syndrome (symptoms occurring at least 3 days per week), including:
   * Postprandial fullness and/or
   * Early satiation 1.1.2 Epigastric pain syndrome (symptoms occurring at least 1 day per week), including:
   * Epigastric pain and/or
   * Epigastric burning 1.2 Participants undergo esophago-gastro duodenoscopy (EGD) to confirm the absence of any structural abnormalities.
2. Control group

   * Patients with no or minimal upper GI symptoms (not match the criteria of FD) and current EGD appear normal or insignificant gastritis
   * Age- and sex-matched to the functional dyspepsia (FD) patient group.

Exclusion Criteria:

* Participants with known organic causes of dyspepsia, including peptic ulcers, gastrointestinal malignancies, or inflammatory bowel disease
* Participants with a history of gastric or hepatobiliary surgery
* Participants who have taken antibiotics and probiotics (as supplements) within 4 weeks before the study
* Participants with significant systemic illnesses, including severe liver or kidney disease, immunodeficiency disorders, or autoimmune diseases
* Pregnant or breastfeeding participants
* Participants who are unable or unwilling to undergo endoscopic procedures for duodenal mucosa collection
* Participants who have taken PPI within 2 weeks before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who were diagnosed with functional dyspepsia according to the ROME IV criteria at King Chulalongkorn Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Specific microbial genus using mucosal brushing | Through study completion, estimated 1.5 years
  The difference of specific duodenal microbiota between patients with functional dyspepsia (FD) and control.
Microbiome diversity using mucosal brushing | Through study completion, estimated 1.5 years
  The difference of specific duodenal microbiome diversity between patients with functional dyspepsia (FD) and control.

SECONDARY OUTCOMES:
Specific microbial genus using mucosal biopsy | Through study completion, estimated 1.5 years
  The difference of specific duodenal microbiota between patients with functional dyspepsia (FD) and control.
Microbiome diversity using mucosal biopsy | Through study completion, estimated 1.5 years
  The difference of specific duodenal microbiome diversity between patients with functional dyspepsia (FD) and control.

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand